CLINICAL TRIAL: NCT01294033
Title: Effect of Therapeutic Hyperoxia on Maximal Oxygen Consumption and Perioperative Risk Stratification in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Supplemental Oxygen on Maximal Oxygen Consumption in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, David H. Roberts, Steven P. Simcox, Patrick A. Clifford and James H. Higby Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2009P000142
Record Dates: First submitted 2011-02-03; First posted 2011-02-11 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fractional inspired oxygen 0.21 (Placebo Comparator): Cardiopulmonary exercise test performed by subject on Fractional inspired oxygen 0.21
  Interventions: Other: Fractional inspired oxygen (FiO2) 0.21
- Fractional inspired oxygen 0.28 (Active Comparator): Cardiopulmonary exercise test performed on supplemental oxygen (Fractional inspired oxygen 0.28)
  Interventions: Other: Fractional inspired oxygen 0.28

INTERVENTIONS:
Other: Fractional inspired oxygen (FiO2) 0.21
  Arms: Fractional inspired oxygen 0.21
Other: Fractional inspired oxygen 0.28 — Supplemental oxygen
  Arms: Fractional inspired oxygen 0.28

SUMMARY:
Maximal consumption of oxygen (VO2max) during exercise is used in patients with chronic obstructive pulmonary disease (COPD) to stratify perioperative risk. However, the impact of supplemental oxygen to prevent hypoxemia during exercise on maximal oxygen consumption and other ventilatory parameters during maximal exercise in the resting normoxic Chronic Obstructive Pulmonary Disease population is poorly defined. The investigators performed a randomized controlled trial in patients with COPD who underwent cardiopulmonary exercise tests on room air and supplemental oxygen. The investigators compared maximal oxygen consumption and other ventilatory parameters in each individual subject under the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD).
* Pulmonary function characterized by forced expiratory volume in 1 second/forced vital capacity ratio<0.7, and forced expiratory volume in one second <80% predicted.

Exclusion Criteria:

* Subjects with a recent COPD exacerbation requiring emergency department visit or hospitalization within the last month.
* Subjects scheduled for a major pulmonary intervention in the next 3 months
* Subjects with severe peripheral vascular disease or other physical conditions that would preclude exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption | Outcomes are measured at time of study visit when patient reaches maximal exercise during cardiopulmonary exercise test. Measurements occur at time of test within 30 minutes of exercise. This is not a longitudinal study measuring outcomes over time.

SECONDARY OUTCOMES:
Minute ventilation - Carbon dioxide production slope | Outcomes are measured at time of study visit when patient reaches maximal exercise during cardiopulmonary exercise test. Measurements occur at time of test within 30 minutes of exercise. This is not a longitudinal study measuring outcomes over time.
Exercise time | Outcomes are measured at time of study visit when patient reaches maximal exercise during cardiopulmonary exercise test. Measurements occur at time of test within 30 minutes of exercise. This is not a longitudinal study measuring outcomes over time.
Oxygen saturation | Outcomes are measured at time of study visit when patient reaches maximal exercise during cardiopulmonary exercise test. Measurements occur at time of test within 30 minutes of exercise. This is not a longitudinal study measuring outcomes over time.
Maximum watts achieved | Outcomes are measured at time of study visit when patient reaches maximal exercise during cardiopulmonary exercise test. Measurements occur at time of test within 30 minutes of exercise. This is not a longitudinal study measuring outcomes over time.
Maximum minute ventilation | Outcomes are measured at time of study visit when patient reaches maximal exercise during cardiopulmonary exercise test. Measurements occur at time of test within 30 minutes of exercise. This is not a longitudinal study measuring outcomes over time.

CONTACTS AND LOCATIONS:
Overall Officials: David H Roberts, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States